CLINICAL TRIAL: NCT05488535
Title: Non-significant Risk Study of a Cochlear Implant Headpiece
Status: Completed | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190256
Record Dates: First submitted 2022-07-26; First posted 2022-08-04 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss; Sensorineural Hearing Loss
Keywords: cochlear implant
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Non-significant risk study of a cochlear implant headpiece (Experimental): This arm aims to evaluate a cochlear implant headpiece.
  Interventions: Device: cochlear implant headpiece

INTERVENTIONS:
Device: cochlear implant headpiece — investigational cochlear implant headpiece

SUMMARY:
This study aims to evaluate a cochlear implant headpiece.

DETAILED DESCRIPTION:
The headpiece and magnet are expected to provide acceptable comfort and retention for existing cochlear implant users. In this study participants will report on their experience with the investigational headpiece during daily life.

ELIGIBILITY:
Inclusion Criteria:

* Pre- or post-lingually deafened.
* Fluent in English, French, or Spanish or capable of communication with a caregiver who is providing consent.
* Adult or child implanted with a commercially available Advanced Bionics cochlear implant. Children and adult participants are included to ensure device retention is appropriate for all implant populations.
* Have (or caregivers have) the cognitive and functional capability to comply with all directions during the study
* Be able to remove their own headpiece
* Have (or caregivers have) the cognitive and functional capability to complete the questionnaire required for the study
* Capable (or caregivers are capable) of reading and understanding patient information materials and giving written informed consent

Exclusion Criteria:

* Have any significant medical condition that, in the opinion of any of the investigators, is likely to interfere with study procedures or likely to confound evaluation of study data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Bionics, Valencia, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Participants eligible to participate in this study were evaluated according to the inclusion requirements for the study. Informed consent was obtained before any study-specific tests or procedures are conducted. An individual was considered to be enrolled as a study participant only after the informed consent document was signed and dated. Each participant was assigned a unique identifier at the time of enrollment. There was only one group of participants for the overall study.
Period: Overall Study
Arm/Group | Overall Study
Started | 101
Completed | 96
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Non-significant Risk Study of a Cochlear Implant Headpiece
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 54
  >=65 years | 41
Age, Continuous [Median (Full Range); unit: years] | 62 [9 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Subjective Report of Headpiece Comfort and Retention
Description: Comfort and subjective retention of the headpiece were rated via questionnaire for baseline headpiece and investigational headpiece acute and chronic use. Subjects were provided with ratings questionnaires and asked to chronically evaluate the headpiece and associated magnet for comfort and retention every two months. Results are presented as total count of participants who rated retention and comfort as favorable ("no opinion," "acceptable," or "very acceptable") at study close out.
  The baseline/investigational headpiece questionnaires included 2 questions:
  1. Rate the retention of your personal/investigational headpiece (Very acceptable, Acceptable, No Opinion, Unacceptable, Very Unacceptable)
  2. Rate the comfort of your personal headpiece (Very acceptable, Acceptable, No Opinion, Unacceptable, Very Unacceptable)
Time Frame: Assessed every two months from month 2 to month 12, values at study close out (month 12) reported.
Population: Subject count at baseline (n=100, includes all subjects enrolled) differ from the overall number of participants analyzed at study close-out (n=72, includes all subjects who were wearing headpiece at the end of the study and who completed final questionnaire).
Measure: Count of Participants; unit: Participants
Arm/Group | Non-significant Risk Study of a Cochlear Implant Headpiece
Number analyzed (Participants) | 72
Participants
  Favorable Retention Rating | 65
  Favorable Comfort Rating | 70

ADVERSE EVENTS:
Time Frame: Issues were reported either by way of direct communications between the trial participants and investigators (verbal, email, phone, etc.) during the active phase of the study (11 months total).
Arm/Group | Non-significant Risk Study of a Cochlear Implant Headpiece
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 2/101
Other Adverse Events (participants affected / at risk) | 5/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-significant Risk Study of a Cochlear Implant Headpiece (N=101)
Skin Flap Thinning Procedure (Surgical and medical procedures) | 2 (2) — The investigational headpiece and magnet were not sufficient in providing acceptable and comfortable retention. Subject had skin flap thinning procedure to ensure headpiece retention was acceptable.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-significant Risk Study of a Cochlear Implant Headpiece (N=101)
Device Temperature (Product Issues) | 1 (1) — Report of investigational device being hot to touch and unwearable. Use of the device was discontinued and returned for analysis, no issue found. No further issues were reported. The issue considered resolved.
Dizziness (Ear and labyrinth disorders) | 1 (1) — Subject reported dizziness when using the investigation device while wearing a headband. After removal of the headband, subject reported feeling dizzy. Subject returned to personal device with a headband. No additional issues were reported.
Headache (General disorders) | 2 (2) — Subject reported experiencing headaches for several months using the investigational device. Subject stopped wearing the investigational device and returned to personal device. Subject reported headaches resolved.
Skin Redness (Skin and subcutaneous tissue disorders) | 1 (1) — Subject self-reported redness of the skin from the investigational device. Site was checked by their audiologist. No redness was reported. The subject continued using the investigational device without incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT05488535/Prot_000.pdf